CLINICAL TRIAL: NCT02964663
Title: Comparison of the Ability of the esCCO and the Volume View to Measure Trends in Cardiac Output During Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Sarah Saxena, MD, Université Libre de Bruxelles
Other Study IDs: EsCCO vs VV
Record Dates: First submitted 2016-11-05; First posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Cardiac Output, Low; Anesthesia
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: esCCO — comparison of non-invasive monitoring esCCO vs VV on cardiac output measurements
  Other Names: VV

SUMMARY:
The purpose of this study was to compare CO measured by two easy to use non-invasive monitors, the esCCO (Nihon Kohden, Tokyo, Japan) to the Volume View (Edwards Lifesciences, Irvine, USA) and to assess their trending ability in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Cardiac output (CO) is a major physiological variable that should be monitored closely during cardiac surgery in order to assess and guide therapeutic interventions so as to decrease postoperative morbidity. The purpose of this study was to compare CO measured by two easy to use non-invasive monitors, the esCCO (Nihon Kohden, Tokyo, Japan) to the Volume View (Edwards Lifesciences, Irvine, USA) and to assess their trending ability in patients undergoing cardiac surgery. After Internal review board approval and written informed consent, 19 patients were included in this study. Before cardiopulmonary bypass (CPB), CO was measured simultaneously using both the esCCO and the Volume View device before and after 3 CO-modifying maneuvers [passive leg raise (PLR), end expiratory occlusion test (EEOT) and positive end expiratory pressure (PEEP) at 10 cm H2O. Five CO values for esCCO and three for volume view were averaged and compared during a one minute period of time before and after each maneuver. The precision error and its 95% confidence interval (CI) that corresponds to the least significant change (LSC) were calculated within this period of time. The Bland-Altman analysis was used to compare bias, precision and limits of agreement (LOA) of both devices. Trending ability of CO changes was assessed by a modified 4 quadrant plot analysis, within angular limits of agreement considered as acceptable when the mean angle between both delta CO was less than 30°.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective cardiac surgery

Exclusion Criteria:

* age less than 18 years
* known or potential pregnancy
* arrhythmias
* known significant tricuspid or aortic valve insufficiency
* left or right ventricular dysfunction
* peripheral arteriopathy
* low perfusion index.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective cardiac surgery
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
interchangeability of both devices (esCCO vs VV) | 6 months
  CO (L/min) was measured using esCCO and VV before and after 3 CO-modifying maneuvers (passive leg raise, PEEP of 10 cmH20, end expiratory occlusion test. Five CO values for esCCO and three for VV were averaged and compared during one minute period of time before and after each maneuver.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasme Hospital, Brussels, Brussels Capital, Belgium